CLINICAL TRIAL: NCT02070263
Title: Mixed Tree Nut Food Challenges
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 110035
Record Dates: First submitted 2013-08-08; First posted 2014-02-25 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Food Allergy
Keywords: Food allergy; Tree nuts
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this prospective study is twofold: 1) to establish oral tolerance to selected tree nuts and to examine potential predictors of oral tolerance and 2) to determine the usefulness of mixed tree nut allergen food challenges in more efficiently defining tree nut allergy and oral tolerance.

DETAILED DESCRIPTION:
To evaluate the absence of tree nuts (TN) allergy, referred patients from one of the Arkansas Children's Hospital (ACH) Allergy Clinic physicians with current serum immunoglobulin E (IgE) to TNs that meet eligibility criteria will be invited to undergo a series of open mixed TN food challenges.

A questionnaire pertaining to their TN allergy will be administered

A brief physical exam will be performed.

Skin prick tests using selected nut allergen extracts along with a positive (histamine) and a negative (salt-water) control will be performed at the first oral food challenge visit.

Each food challenges will be performed to 1 to 3 TNs.

Two telephone follow-up phone calls will evaluate inclusion/exclusion of tree nuts in the diet post food challenge.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between 3-21 years of age followed by the Allergy and Immunology Department at Arkansas Children's Hospital on tree nut avoidance diet.
* Has current serum IgE test within the past 12 months to major nuts in question. All TN serum IgE are <10
* Children must have a stable baseline examination prior to undergoing challenge without significant symptoms of atopic dermatitis, allergic rhinoconjunctivitis, current urticaria or other allergic symptoms deemed important by the physician.
* Children must have stable asthma and no wheezing or repetitive cough prior to challenge, nor have been treated with oral steroids for a significant asthma exacerbation within 1 month of challenge. Asthmatics that undergo lung function testing.
* Children must have no current illness (e.g., fever or viral illness) at time of challenge.
* The subject will be asked to restrict the use of antihistamines (short acting, 72 hours: long acting, 5-7 days), (B-agonists (12 hours), theophylline (12 hours), and cromolyn (12 hours) prior to the first mixed TN food challenge. Other medications may be continued.

Exclusion Criteria:

* Any TN serum IgE ≥10.
* Life-threatening reaction (respiratory involvement requiring medications, or shock, or gastrointestinal reaction requiring intravenous fluids) to any TN.
* History of a reaction in the past year or severe reaction in the past 2 years or a history of a severe reaction anytime with a TN serum IgE >5
* Unstable asthma, gastrointestinal disease, cardiovascular disease, chronic lung disease, beta-blocker use.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients seen at Arkansas Children's Hospital between 3-21 years of age who have tree nut food allergies.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Oral tolerance to selected tree nuts (TN) to determine potential predictors of oral tolerance. | total -20 years
  This prospective, observational study uses serum IgE to specific TN, skin prick test to TN, and TN oral food challenges to establish oral tolerance.

SECONDARY OUTCOMES:
Use of tree nut (TN) IgE testing to assess the risk of positive food challenges based on grouped mixed TN food challenges | total - 20 years
  We postulate that by grouping TN that are mixed into one food challenge based on the individual's TN serum IgE will be more efficient in defining TN allergy and tolerance. One to three TNs will be in one food challenge based on TN IgE testing.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie M Jones, MD, Principal Investigator — University of Arkansas for Medical Sciences / Arkansas Children's Hospital
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data has not been analyzed at thistime